CLINICAL TRIAL: NCT03240913
Title: A PROMs Based Educational Tool (PROM-DA) for Patients Considering Total Knee Arthroplasty: Development and a Pilot Randomized Controlled Trial.
Brief Title: A PROMs Based Educational Tool (PROM-DA) for Patients Considering Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB16-0869
Record Dates: First submitted 2017-07-27; First posted 2017-08-07 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental)
  Interventions: Behavioral: Baseline and Follow-up Surveys; Other: Patient Reported Outcome Measure informed Decision Aid
- Non Treatment Group (Placebo Comparator): Conventional information
  Interventions: Behavioral: Baseline and Follow-up Surveys; Other: Pamphlet

INTERVENTIONS:
Behavioral: Baseline and Follow-up Surveys — (completed online)
Other: Patient Reported Outcome Measure informed Decision Aid — (PROM-DA)
  Arms: Treatment Group
Other: Pamphlet — (usual care)
  Arms: Non Treatment Group

SUMMARY:
The primary objectives of this study are to: 1) develop an educational tool known as the Patient Reported Outcome Measure informed Decision Aid (PROM-DA) that will describe the options for patients considering total knee arthroplasty (TKA) surgery, and help them imagine what to expect if they choose either option; 2) assess the extent that the PROM-DA improves patients decision quality; 3) determine the feasibility of a larger trial to test the PROM-DA in multiple sites and more patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age≥30) patients with knee osteoarthritis (OA)
* Have an appointment with a surgeon for consultation about Total Knee Arthroplasty at the Edmonton Bone and Joint Centre
* Understands, speaks and reads English; and
* Able to provide informed consent.

Exclusion Criteria:

* Individuals who have had prior total knee arthroplasty
* Physician-diagnosed Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis, Fibromyalgia, or Gout.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Decision quality | 40 to 52 weeks after baseline
  Hip and Knee Decision Quality Instrument (HK-DQI)

SECONDARY OUTCOMES:
Quality of life (generic) | 40 to 52 weeks after baseline
  Euroqol Five Dimensions Questionnaire (EQ-5D-5L)
Quality of life (condition-specific) | 40 to 52 weeks after baseline
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Depression | 40 to 52 weeks after baseline
  The Patient Health Questionnaire (PHQ-9)
Knowledge about total knee arthroplasty surgery | Baseline
  HK-DQI
Values | Baseline
  HK-DQI
Decisional conflict | Baseline
  Decisional Conflict Scale (SURE)
Treatment Preference | Baseline
  Single item question: Do you feel the potential benefits of knee replacement surgery outweigh the potential surgical risks?
  Yes No Unsure
Preference for involvement in decision making | Baseline
  Control Preferences Scale (CPS)
Willingness to have surgery | Baseline
  Single item question: Based on your current understanding of the risks and benefits of knee replacement surgery of your knee arthritis, what is your current preference between having joint replacement surgery or non-surgical treatments?
  I would definitely consider having knee joint replacement surgery now. I would probably consider having knee joint replacement surgery now. I am not sure. I would probably not consider having knee joint replacement surgery now. I would definitely not consider having knee joint replacement surgery now.
Patient-reported shared decision-making | 3 to 6 weeks after baseline
  CollaboRATE
Decisional regret | 40 to 52 weeks after baseline
  Decision Regret Scale
Satisfaction with knee replacement surgery | 40 to 52 weeks after baseline
  Three item questionnaire:
  1. Overall, how satisfied are you with the results of your knee replacement surgery?
  2. How satisfied are you with your knee replacement surgery for reducing your pain when walking on a flat surface? Going up or down stairs? Sitting or lying down?
  3. How satisfied are you with your most recent knee replacement surgery for improving your ability to perform five functions: Going up stairs? Getting in/out of a car or on/off a bus? Rising from bed? Lying in bed? Performing light domestic duties?
  Responses from 'very dissatisfied' to ' very satisfied'
Expectations | 40 to 52 weeks after baseline
  Single item question from Bourne et al. 2010. Clin Orthop Relat Res. related to whether expectations were met; not met; or whether they had no expectations.
Surgical consult | 1 to 4 weeks after baseline
  Electronic Medical Records (EMR)
Surgery | 27 to 30 weeks after baseline
  EMR
Concordance | 40 to 52 weeks after baseline
  HK-DQI

CONTACTS AND LOCATIONS:
Locations (1):
- Edmonton Bone and Joint Centre, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bansback N, Trenaman L, MacDonald KV, Hawker G, Johnson JA, Stacey D, Marshall DA. An individualized patient-reported outcome measure (PROM) based patient decision aid and surgeon report for patients considering total knee arthroplasty: protocol for a pragmatic randomized controlled trial. BMC Musculoskelet Disord. 2019 Feb 23;20(1):89. doi: 10.1186/s12891-019-2434-2. PMID 30797238